CLINICAL TRIAL: NCT06409923
Title: Comparison of Skeletal Effects of Herbst and Invisalign MA in Growing Patients With KLass Malocclusion
Brief Title: Comparison of Skeletal Effects of Herbst and Invisalign MA in Growing Patients With KLass II Malocclusion
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Paul-Henry Casselman, Postgraduate student Dentofacial orthopedics and orthodontics, Université Libre de Bruxelles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRB2023175
Record Dates: First submitted 2024-04-09; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Mandibular Growth Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Invisalign MA- group (mandibular advancement) (Active Comparator): Patients treated by MA aligner system of invisalign
  Interventions: Device: Stimulation of mandibular growth.
- Herbst group (Active Comparator): Patient treated with the herbst appliance
  Interventions: Device: Stimulation of mandibular growth.

INTERVENTIONS:
Device: Stimulation of mandibular growth. — orthodontic treatment where a retrognathic mandibula is put into an anterior position to stimulate mandibular growth. This will happen by either the MA-invisalign system or the herbst appliance

SUMMARY:
This study aims to determine and compare the precise skeletal dental and soft tissue effect of Mandibular advancement aligners and Herbst Appliance.

DETAILED DESCRIPTION:
Precise description of study methodology.

For each group, a sample of +- 15 patients with class 2 malocclusion aged between 9 and 15 years will be collected for this prospective study who presented for an initial orthodontic consultation between October 2022 and july 20262 at ULB's Erasme Hospital. Each patient will be treated with Invisalign MA or the Herbst appliance by residents of the orthodontic program directed by P. Maria Orellana

Inclusion criteria included a Class II skeletal malocclusion with an ANB greater than 4°; (In the case of a Class 2 Division 2 malocclusion, the retroclined upper incisors will be proclined to obtain an overjet allowing mandibular advancement. If the patient has a transverse deficit, palatal expansion will be performed before treatment with aligners and during treatment in herbst cases.) Class II molar and canine relationship and CVM2/CVM3 cervical vertebral maturation.

Informed consent forms in the patient's native language will be submitted before the start of each treatment.

Only a profile cephalometry will be taken in the patients considered for this study at the time of the initial consultation.

This will avoid unnecessary radiographic exposure, and a panoramic view of each patient will be extracted from a CBCT using the FDA-approved BlueskyBio program.

Aligners or Herbst appliance for orthodontic treatment will be fabricated on the basis of a 3D optical scan (Itero), after which patients will begin treatment.

Levelling of the Spee curve, derotation of (pre)molars and palatal incisors in the case of class 2 division 2 malocclusion will be carried out before the mandibular advancement stage if necessary in the Aligner group.

A full-face ultra-low dose CBCT scan will be performed on all included subjects before the mandibular advancement stage according to a strict protocol by a certified physician. Active mandibular advancement will be continued till a KLass I molar relationship is obtained and will be followed by 2 months without mandibular advancement to allow the mandibular condyles to take a central position in the condylar fossae. After this 2-month period, a second CBCT scan will be performed (T2), with a minimal time interval of one year between the two CBCT scans, using the same protocol.

CBCTs will be acquired using a Promax Mid 90 Kv with settings of 90 kV and 8.9 mAS, and tube current modulation will be used to enable patient-specific dose reduction.

After the second CBCT, orthodontic treatment will be continued until completion, and retention and regular post-treatment follow-up will be scheduled for each patient.

The superposition of CBCT (T1) and (T2) images on the anterior cranial base will be used to determine exact mandibular lengthening, condylar displacement, mandibular rotation and chin displacement using the following methodology described and developed by Hugo. De Clerck in 2009.

ELIGIBILITY:
Inclusion Criteria

* ANB greater than 4°.
* Angle Class II molar and canine relationship
* cervical vertebral maturation (CVM) CVM2/CVM3

Exclusion Criteria:

* CVM> 4
* periodontal disease

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2027-09-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Mandibular lenghtening | Difference between T1/T2. T1: Before Mandibular advancement phase, T2: Minimum 1 year after T1 and 2 months without mandibular advancement.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Université LIbre de Bruxelles, Anderlecht
  - UNiversité Libre de Bruxelles, Brussels

IPD SHARING:
Plan to Share IPD: No